CLINICAL TRIAL: NCT05841173
Title: Effects of Weight Loss Management on Cognitive Function in Elderly Obese Women
Brief Title: Effects of Weight Loss Management on Cognitive Function in Elderly Women With Obesity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal State Budgetary Scientific Institution "Federal Research Centre of Nutrition, Biotechnology (Other)
Collaborators: Federal Stare Budgetary Scientific Institution, Mental Health Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: ВОВ-01
Record Dates: First submitted 2023-04-10; First posted 2023-05-03 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Obesity; Cognitive Change
Keywords: Elderly; Obesity; Weight loss; Cognitive Change; Exogenous Ketones; Diet; Physical activity
MeSH Terms: conditions — Obesity; Weight Loss; Motor Activity | interventions — Exercise; Diet

STUDY DESIGN:
Intervention Model Description: Prospective randomised parallel arms double control interventional study
Who Masked: Participant, Investigator
Masking Description: Masking is used between 2 groups out of 5 (between the Product group and Placebo group). The investigated product and Placebo have comparable organoleptic properties and are packed in the same containers labelled as N1 or N2.
  The participants are randomised for 5 arms. In the case of arms 1 and 2, they are prescribed to consume 2 doses of product per day without awareness of either it is the investigational product or a placebo (the investigational product or a placebo). Field investigators prescribe to participants product N1 or N2 according to group allocation without awareness of either it is the investigational product or a placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- The Product Group (Experimental): The Product group is prescribed with the investigated product - exogeneous ketone bodies.
  Interventions: Dietary Supplement: "PanTrek"
- The Combined Intervention Group (Active Comparator): The Combined Intervention Group is prescribed with the investigated product -in combination with regular physical trainings.
  Interventions: Dietary Supplement: "PanTrek"; Behavioral: Physical Trainings
- The Placebo Group (Placebo Comparator): The Placebo Group is prescribed with the Placebo.
  Interventions: Other: Placebo
- The Diet Group (Active Comparator): The Diet Group is prescribed with the Diet designed with 500 kcal reduction from daily energy expenditure.
  Interventions: Behavioral: Diet
- The Control Group (No Intervention): The Control Group is prescribed with standard recommendations for weight loss.

INTERVENTIONS:
Dietary Supplement: "PanTrek" — The intervention is represented by the investigational product "PanTrek", shots with liquid, 25 ml each (TU 10.89.19-01-44850857-2020). The composition of the product "PanTrek" (per 1 dose):
  * Ginseng dry extract (Panax ginseng Meyer) all parts of the plant - 125 mg (the amount of ginsenosides in one vial is 9.0 mg ± 3.5 mg);
  * Melissa officinalis dry extract (Melissa officinalis L) all parts of the plant - 340 mg (the amount of hydroxycinnamic acids is 19.50 mg / vial ± 10% in one vial);
  * Apple juice concentrated 2.5% - 7,5 g;
  * Potassium beta-hydroxybutyrate - 4,5 g;
  * Magnesium beta-hydroxybutyrate - 500 mg;
  * E211 sodium benzoate - no more than 5 mg;
  * E202 Potassium sorbate - no more than 3,6 mg;
  * Water purified - up to 25 ml. The product has registered as diet supplement in the Unified Register of Certificates of State Registration N RU.77.99.11.003.R.001152.04.21 from 05.04.2021.
  Other Names: Exogenous ketone bodies
  Arms: The Combined Intervention Group; The Product Group
Behavioral: Physical Trainings — Physical activity is represented by 2 workouts lasting 45 minutes per week on an antigravity treadmill Alter-G M320 (AlterG, USA) and 2 sessions of reoxygenation lasting 30 minutes on a normobaric hypoxic therapy device ReOxy (Bitmos GmbH, Germany).
  Other Names: Exercises
  Arms: The Combined Intervention Group
Other: Placebo — The placebo is represented by concentrated apple juice 2.5% - 7.5 g, potassium chloride - 2.405 g, MgCl2 - 0.382 g, sodium benzoate (E211) - 5 mg and potassium sorbate (E202) - 3.6 mg, brought to 25 ml of distilled water.
  Arms: The Placebo Group
Behavioral: Diet — The studied diet is a low-calorie diet with an average energy value of 1730.16 kcal / day and a certain chemical composition (proteins - 108.80 g / day, fats - 68.10 g / day, carbohydrates - 162.60 g / day), including the main groups products (meat and poultry dishes, fish dishes, dairy products, cereals, vegetables and fruits). On average, 0.96-1.05 g of protein accounted for 1 kg of body weight of the subjects.
  Arms: The Diet Group

SUMMARY:
According to studies, the risk of cerebrovascular disease and cognitive decline are associated with age-related changes. In addition, there is data suggesting a relationship between the progression of this pathology and the presence of obesity and associated metabolic disorders. According to to some research, weight loss associated with cognitive function decline. In this regard, the development of effective, applicable in real clinical practice methods of non-drug treatment and prevention of cerebrovascular disorders and age-related cognitive decline in people with obesity and metabolic disorders, who are at high risk, seems to be extremely relevant.

The main goal of the study is to compare the effectiveness of various weight loss approaches and to study their effects on the cognitive functions of elderly obesity women.

DETAILED DESCRIPTION:
The high prevalence of comorbid pathology characterised the elderly and senile population. Particularly, comorbid condition is often based on obesity. Also, an important characteristic of the elderly and senile age is the development of age-related cognitive deficit and progressive decline in cognitive functions, that is detected in 60.8% of people over 65 years old in Russia according to the EVKALIPT study.

The prevalence of obesity in the Russian population reaches 40% among the elderly population. According to studies, the presence of obesity is "paradoxically" associated with less progression of cognitive function loss, and the risk reduction in some populations reaches 40%. However, the sarcopenic obesity is an independent predictor of cognitive impairment in the elderly. Consequently, the therapy of obesity in elderly and senile population faces two important aspects: the risk of muscle loss and the development of sarcopenia and progressive cognitive decline. The described features of this age group are consistent with the well-known "obesity paradox", in which overweight and obesity are associated with longer life expectancy.

The risk of muscle mass reduction and cognitive functions decrease determines the formation of a specialised approach to obesity management in older population. Thus, the setting of softer and longer-term goals with a gradual decrease in body weight is typical. Studies have considered the use of various interventions, so far the combination of diet with exercise has proven effectiveness in muscle mass protection. At the same time, regular exercises reliably protect from cognitive decline. Thereby, the combination of diet and physical activity is considered as a suitable approach to obesity management in the elderly.

Recently, there have also been a number of studies evaluating the effectiveness of the ketogenic diet. This diet pattern is reliably effective in body weight reduction, skeletal muscle mass maintenance, and adipose tissue metabolism improvement in the elderly . Also, the neuroprotective effects of the ketogenic diet have been confirmed by meta-analyses and have made it possible to include it in current guidelines for the prevention and treatment of cognitive impairment. However, the high frequency of negative effects and the associated low adherence limit the possibilities of using this diet, which led to the development of exogenous ketones that allow reaching the levels of blood ketone bodies associated with neuroprotective properties (0.2-0.5 mmol/l) with better portability.

The main goal of the study is to compare the effectiveness of various weight loss approaches and to study their effects on the cognitive functions of elderly obesity women.

ELIGIBILITY:
Inclusion Criteria:

1. Female;
2. Age 60 and over;
3. BMI 30.0 kg/m2 or more.

Exclusion Criteria:

1. Male;
2. age under 60;
3. BMI <30.0 kg/m2;
4. patients unable or unwilling to comply with the requirements of the protocol, including the signing of informed consent (inability to give such consent due to mental deficiency or language barrier), as well as non-compliance with the schedule of visits, persons unable to independently make a decision and sign an informed consent;
5. less than 6 months after suffering cardiovascular events, stroke, severe surgical interventions and injuries;
6. alcohol abuse (including chronic pancreatitis of alcoholic etiology) or drug addiction at present or within the last 5 years;
7. history of malignant diseases, regardless of the treatment during the last 5 years;
8. less than 4 weeks after suffering acute infectious and / or inflammatory diseases, after the onset of complete clinical and laboratory remission;
9. pregnancy and lactation;
10. history of allergic reactions to components of the study product and/or placebo or intolerance to components of the study product and/or placebo.

Ages: 60 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The females participants are reqruited In order to reduce variability of results in the restricted sample size (40 person per group).
Enrollment: 200 (Estimated)
Dates: Start 2022-01-09 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline body weight at 12 weeks | Baseline (visit 1) and after 12 weeks (visit 2)
  The dynamics of body weight
Change from baseline Montreal Cognitive Assessment (MoCa) test scores at 12 weeks | Baseline (visit 1) and after 12 weeks (visit 2)
  The changes in the cognitive testing results
Change from baseline Trail Making Test (TMT) a&b test scores at 12 weeks | Baseline (visit 1) and after 12 weeks (visit 2)
  The changes in the cognitive testing results (normal range - less than 78 and 273 seconds (=scores)).
Change from baseline Word recall test scores at 12 weeks | Baseline (visit 1) and after 12 weeks (visit 2)
  The changes in the cognitive testing results (normal range as 45 words (=scores) and more out of 5 repetitions). Minimal - 0 (worse result), maximal score - 50 (excellent result).
Change from baseline Mean response time in the test "Schulte tables" at 12 weeks | Baseline (visit 1) and after 12 weeks (visit 2)
  The changes in the cognitive testing results
Change from baseline The Stroop Color and Word Test results at 12 weeks | Baseline (visit 1) and after 12 weeks (visit 2)
  The changes in the cognitive testing results
Change from baseline Verbal fluency test results at 12 weeks | Baseline (visit 1) and after 12 weeks (visit 2)
  The changes in the cognitive testing results

SECONDARY OUTCOMES:
Change from baseline fat mass at 12 weeks | Baseline (visit 1) and after 12 weeks (visit 2)
  The changes in the fat mass according to the bioimpedance analysis
Change from baseline skeletal muscle mass at 12 weeks | Baseline (visit 1) and after 12 weeks (visit 2)
  The changes in the skeletal muscle mass according to the bioimpedance analysis
Change from baseline visceral fat at 12 weeks | Baseline (visit 1) and after 12 weeks (visit 2)
  The changes in visceral fat according to the bioimpedance analysis
Change from baseline total cholesterol serum levels at 12 weeks | Baseline (visit 1) and after 12 weeks (visit 2)
  The changes of total cholesterol serum levels
Change from baseline LDL-cholesterol serum levels at 12 weeks | Baseline (visit 1) and after 12 weeks (visit 2)
  The changes of LDL-cholesterol serum levels
Change from baseline HOMA-IR (homeostasis model assessment - insulin resistance) index at 12 weeks | Baseline (visit 1) and after 12 weeks (visit 2)
  The changes of HOMA-IR index
Change from baseline C-reactive protein (CRP) serum levels at 12 weeks | Baseline (visit 1) and after 12 weeks (visit 2)
  The changes of CRP serum levels
Change from baseline Tumor Necrosis Factor Alpha (TNFa) serum levels at 12 weeks | Baseline (visit 1) and after 12 weeks (visit 2)
  The changes of TNFa serum levels
Change from baseline systolic blood pressure (SBP) at 12 weeks | Baseline (visit 1) and after 12 weeks (visit 2)
  The changes of SBP
Change from baseline diastolic blood pressure (DBP) at 12 weeks | Baseline (visit 1) and after 12 weeks (visit 2)
  The changes of DBP
Change from baseline grip strength at 12 weeks | Baseline (visit 1) and after 12 weeks (visit 2)
  The changes of grip strength measured by grip dynamometer on the leading hand
Change from baseline Six Minute Walk Test distance at 12 weeks | Baseline (visit 1) and after 12 weeks (visit 2)
  The changes of Six Minute Walk Test results
Change from baseline Hamilton Anxiety Rating Scale at 12 weeks | Baseline (visit 1) and after 12 weeks (visit 2)
  The changes of Hamilton Anxiety Rating Scale results (normal range - 6 scores and less).
Change from baseline Hamilton Depression Rating Scale at 12 weeks | Baseline (visit 1) and after 12 weeks (visit 2)
  The changes of Hamilton Depression Rating Scale results (normal range - 7 scores and less).

CONTACTS AND LOCATIONS:
Overall Officials: Antonina V. Starodubova, MD, Full PhD, Study Director — Deputy Director of the Federal Research Centre of Nutrition, Biotechnology and Food Safety; Yurgita R. Varaeva, MD, MRes, Principal Investigator — Research Fellow of the Federal research Centre of Nutrition, Biotechnology and Food Safety
Locations (1):
- Nutrition Clinic of the Federal Research Centre of Nutrition, Biotechnology and Food Safety, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dadarlat-Pop A, Sitar-Taut A, Zdrenghea D, Caloian B, Tomoaia R, Pop D, Buzoianu A. Profile of Obesity and Comorbidities in Elderly Patients with Heart Failure. Clin Interv Aging. 2020 Apr 21;15:547-556. doi: 10.2147/CIA.S248158. eCollection 2020. PMID 32368021
- [Background] Abdoli N, Salari N, Darvishi N, Jafarpour S, Solaymani M, Mohammadi M, Shohaimi S. The global prevalence of major depressive disorder (MDD) among the elderly: A systematic review and meta-analysis. Neurosci Biobehav Rev. 2022 Jan;132:1067-1073. doi: 10.1016/j.neubiorev.2021.10.041. Epub 2021 Nov 4. PMID 34742925
- [Background] Khovasova NO, Vorobyeva NM, Tkacheva ON, Kotovskaya YV, Naumov AV, Selezneva EV, Ovcharova LN. [The prevalence of anemia and its associations with other geriatric syndromes in subjects over 65 years old: data of Russian epidemiological study EVKALIPT]. Ter Arkh. 2022 Jan 15;94(1):24-31. doi: 10.26442/00403660.2022.01.201316. Russian. PMID 36286917
- [Background] Martinchik AN, Laikam KE, Kozyreva NA, Keshabyants EE, Mikhailov NA, Baturin AK, Smirnova EA. [The prevalence of obesity in various socio-demographic groups of the population of Russia]. Vopr Pitan. 2021;90(3):67-76. doi: 10.33029/0042-8833-2021-90-3-67-76. Epub 2021 May 17. Russian. PMID 34264558
- [Background] Hou Q, Guan Y, Yu W, Liu X, Wu L, Xiao M, Lu Y. Associations between obesity and cognitive impairment in the Chinese elderly: an observational study. Clin Interv Aging. 2019 Feb 15;14:367-373. doi: 10.2147/CIA.S192050. eCollection 2019. PMID 30863030
- [Background] Vidyanti AN, Hardhantyo M, Wiratama BS, Prodjohardjono A, Hu CJ. Obesity Is Less Frequently Associated with Cognitive Impairment in Elderly Individuals: A Cross-Sectional Study in Yogyakarta, Indonesia. Nutrients. 2020 Jan 30;12(2):367. doi: 10.3390/nu12020367. PMID 32019161
- [Background] Wang H, Hai S, Liu YX, Cao L, Liu Y, Liu P, Yang Y, Dong BR. Associations between Sarcopenic Obesity and Cognitive Impairment in Elderly Chinese Community-Dwelling Individuals. J Nutr Health Aging. 2019;23(1):14-20. doi: 10.1007/s12603-018-1088-3. PMID 30569063
- [Background] Colleluori G, Villareal DT. Aging, obesity, sarcopenia and the effect of diet and exercise intervention. Exp Gerontol. 2021 Nov;155:111561. doi: 10.1016/j.exger.2021.111561. Epub 2021 Sep 23. PMID 34562568
- [Background] Kokkinidis DG, Armstrong EJ, Giri J. Balancing Weight Loss and Sarcopenia in Elderly Patients With Peripheral Artery Disease. J Am Heart Assoc. 2019 Jul 2;8(13):e013200. doi: 10.1161/JAHA.119.013200. Epub 2019 Jun 29. PMID 31257976
- [Background] Giudici KV, Guyonnet S, Rolland Y, Vellas B, de Souto Barreto P, Nourhashemi F; MAPT/DSA Group. Body Weight Variation Patterns as Predictors of Cognitive Decline over a 5 Year Follow-Up among Community-Dwelling Elderly (MAPT Study). Nutrients. 2019 Jun 18;11(6):1371. doi: 10.3390/nu11061371. PMID 31216732
- [Background] Bosello O, Vanzo A. Obesity paradox and aging. Eat Weight Disord. 2021 Feb;26(1):27-35. doi: 10.1007/s40519-019-00815-4. Epub 2019 Dec 21. PMID 31865598
- [Background] Semlitsch T, Stigler FL, Jeitler K, Horvath K, Siebenhofer A. Management of overweight and obesity in primary care-A systematic overview of international evidence-based guidelines. Obes Rev. 2019 Sep;20(9):1218-1230. doi: 10.1111/obr.12889. Epub 2019 Jul 8. PMID 31286668
- [Background] Petroni ML, Caletti MT, Dalle Grave R, Bazzocchi A, Aparisi Gomez MP, Marchesini G. Prevention and Treatment of Sarcopenic Obesity in Women. Nutrients. 2019 Jun 8;11(6):1302. doi: 10.3390/nu11061302. PMID 31181771
- [Background] Falck RS, Davis JC, Best JR, Crockett RA, Liu-Ambrose T. Impact of exercise training on physical and cognitive function among older adults: a systematic review and meta-analysis. Neurobiol Aging. 2019 Jul;79:119-130. doi: 10.1016/j.neurobiolaging.2019.03.007. Epub 2019 Mar 26. PMID 31051329
- [Background] Ilyas Z, Perna S, A Alalwan T, Zahid MN, Spadaccini D, Gasparri C, Peroni G, Faragli A, Alogna A, La Porta E, Ali Redha A, Negro M, Cerullo G, D'Antona G, Rondanelli M. The Ketogenic Diet: Is It an Answer for Sarcopenic Obesity? Nutrients. 2022 Jan 30;14(3):620. doi: 10.3390/nu14030620. PMID 35276979
- [Background] Buckinx F, Aubertin-Leheudre M. Nutrition to Prevent or Treat Cognitive Impairment in Older Adults: A GRADE Recommendation. J Prev Alzheimers Dis. 2021;8(1):110-116. doi: 10.14283/jpad.2020.40. PMID 33336232
- [Background] McDonald TJW, Cervenka MC. Lessons learned from recent clinical trials of ketogenic diet therapies in adults. Curr Opin Clin Nutr Metab Care. 2019 Nov;22(6):418-424. doi: 10.1097/MCO.0000000000000596. PMID 31503023